CLINICAL TRIAL: NCT03225794
Title: Epidemiological and Molecular Aspects of the Interspecies Transmission of Foamy Viruses From Monkeys to Humans: A Model of the Early Stages of Viral Emergence.
Brief Title: Simian Foamy Virus Transmission to Humans
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010-27
Record Dates: First submitted 2017-07-07; First posted 2017-07-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Simian Foamy Virus Infection (Disorder)
Keywords: Retrovirus; Viral emergence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood draw into a 5/10 ml EDTA tubes; Oral specimens will be collected by rubbing the inside of the cheek with a swab and then rinsing the mouth and collecting the rinse liquid in a sterile bottle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Adults living in rural area of Cameroon, not infected with simian foamy viruses
  Interventions: Diagnostic Test: Simian foamy virus Infection
- Simian Foamy virus infection: Adults living in rural area of Cameroon, infected with simian foamy viruses
  Interventions: Diagnostic Test: Simian foamy virus Infection

INTERVENTIONS:
Diagnostic Test: Simian foamy virus Infection — Plasma samples are tested for the presence of antibodies directed against foamy viruses by western blotting (WB). The BHK-21 cell line infected with a chimpanzee foamy virus is used as a source of viral antigen. Samples are considered to be positive if there is net reactivity against the GAG doublet (70 to 74 kD). High molecular weight DNA will be extracted, from either buffy coats, cell cultures, or both, for molecular biology studies. The presence and quality of the DNA will be verified by amplification of a fragment of the beta-globin gene. Two regions of foamy virus genomic DNA will be amplified by nested PCR, using generic amplimers, giving rise to fragments of the integrase gene (425 bp) and LTR (109 bp).

SUMMARY:
About three quarters of the viral agents that have emerged recently in humans are considered to originate from other animals. These viruses have often evolved and spread into the human population through various mechanisms after the initial contact that resulted in interspecies transmission. However, knowledge of the initial stages of the emergence of viruses and associated diseases is still limited in many cases. Microbiological monitoring in populations at risk of transmission would provide insights into the initiation and early stages of the emergence process.

Nonhuman primates (NHPs) share many genetic, physiological, and microbiological features with humans, and are potential sources of many infectious agents. This has been demonstrated for several simian retroviruses. HIV-1 and 2 are believed to have originated from chimpanzee and mangabey viruses, respectively, found in Central and West Africa. The current distribution of the various molecular subtypes of the HTLV-1 oncogenic retrovirus in Africa is mainly the result of numerous instances of interspecies transmission of STLV-1from NHP species in the distant past.

Foamy viruses belong to the Retrovidae family and the Spumavirus genus. They are complex exogenous retroviruses and are very common in many animal species, including primates, cats, cattle, and horses, in which they cause persistent infections.

The first aim of the work is to study the epidemiological and molecular aspects of the transmission of foamy viruses from monkeys to humans in populations at risk, such as the inhabitants (especially hunters) in the villages of the dense forests of southern Cameroon. It is an area in which NHPs are still very common, with a great diversity of species. The investigators have already shown that the prevalence of foamy viruses is very high in these monkeys and great apes (gorillas and chimpanzees). Contact between these monkeys and the villagers is very frequent, mainly during hunting. The second aim of the project is to study the clinical and biological features of infected people and investigate intrafamilial transmission from infected index cases.

DETAILED DESCRIPTION:
BACKGROUND A large proportion, about 75%, of the viral agents that have emerged recently in humans have originated from other animals. Following the initial contact resulting in interspecies transmission, these viruses have often evolved and spread through the human population; various mechanisms are involved, but the understanding of the initial stages of the emergence of viruses and associated diseases is still limited in many cases.

Microbiological monitoring in populations at risk of transmission is required to identify and document the initiation and early stages of the emergence process.

Nonhuman primates (NPHs), which share many genetic, physiological, and microbiological similarities with humans, are a potential source of many infectious agents.

This has been clearly demonstrated for several simian retroviruses: HIV-1 and 2 are believed to have originated from chimpanzee and mangabey viruses, respectively, in Central and West Africa. The distribution of the various molecular subtypes of the oncogenic retrovirus HTLV-1 in Africa is mainly the result of the pattern of interspecies transmission of STLV-1 from various NHP species in the distant past.

Foamy viruses belong to the retrovidae family and the spumavirus genus. They are complex exogenous retroviruses and are very common in many animal species, including primates, cats, cattle, and horses, in which they cause persistent infections.

Foamy viruses are generally non-pathogenic, even in experimentally infected animals. They do not appear to cause disease in the few humans who have been accidentally infected and clinically and biologically followed-up long-term (fewer than 15 people have been followed to date and they were originally healthy such that there is a selection bias). The absence of pathogenicity in vivo contrasts with the strong cytopathogenic effects of foamy virus in vitro where they cause syncytia in cell cultures.

Unlike lentiviruses (HIV-SIV), foamy viruses are extremely genetically stable in vivo. Phylogenetic analysis has demonstrated genetic variability, depending on the animal species infected. This indicates long coevolution of these retroviruses with their natural hosts. Switzer et al., showed that foamy viruses have coevolved with old world primates for at least 30 million years (Switzer et al. 2005). These data may explain the apparent absence of pathogenicity in vivo despite chronic infection.

The molecular characteristics of foamy viruses have been extensively studied in vitro, but little is currently known about the characteristics of these viruses in vivo, and in particular, about the epidemiological determinants of infection. Indeed, the modes of contamination and the characteristics of the primary infection in humans under natural conditions are still poorly understood.

The rare epidemiological data published are mostly for populations of captive NHPs: the seroprevalence of foamy viruses can reach 75% or more in adults in these populations. Several studies have shown that the saliva of infected animals has high titers of the virus, suggestive of the mode of transmission. The mucosa of the oropharynx is an important site of replication in green monkeys and a recent article reports high levels of viral RNA in saliva and oropharyngeal specimens from macaques. These observations suggest that bites or contact with oral mucosa and saliva can be transmission mechanisms, at least in some cases. Other studies in colonies of captive baboons suggest that transmission can be sexual and/or from mother to child through repeated salivary contact.

Human infection with foamy viruses has been reported: 1 to 4% of people professionally exposed to NHP (such as veterinarians, and personnel who work in animal houses, zoos, and primatology laboratories) in North America and, more rarely, in Europe may be infected.

An American group has shown infection by foamy viruses, originating from gorillas and mandrills, in some hunters living in Cameroon (Wolfe et al. 2004). Some cases of infection have been demonstrated in people in Southeast Asia in contact with monkeys (especially macaques): people working in temples, especially in Indonesia, or involved in hunting or other activities that put them in close contact with monkeys. Mathematical models have estimated that approximately six per 1000 temple visitors in Bali, Indonesia, where there are many macaques, have been infected with a simian foamy virus (Engel et al. 2006).

The long-term collaboration betwwen the investigators, the Pasteur Center of Cameroon, the IRD, and the University of Yaounde I, using serological and molecular techniques (PCR), has demonstrated foamy viruses in wild populations of gorillas, chimpanzees, mandrills, and drills in Cameroon. Adult populations of NHPs in these regions are highly infected with foamy viruses, with a specific virus for each species (Calattini et al. 2004 , Calattini et al. 2006b).

Consistent with the American study cited above, the investigators have demonstrated infection of hunters by the foamy viruses found in gorillas, chimpanzees, and mandrills after having been in contact with these primates (Calattini et al. 2007).

The EPVO unit at Institut Pasteur has been working in close collaboration with the Pasteur Center of Cameroon and the IRD for more than 15 years on numerous epidemiological studies in the field of the human retroviruses HTLV-1 (Mahieux et al. 2000b, Mauclere et al. 1997), HTLV-2(Gessain et al. 1995, Mauclere et al. 1995), the simian retroviruses STLV-1 and STLV-3 (Mahieux et al. 2000a, Meertens et al. 2002, Meertens et al. 2001, Meertens et al. 2003, Nerrienet et al. 2004, Nerrienet et al. 2001), and HTLV-3 (Calattini et al. 2009, Calattini et al. 2006a, Calattini et al. 2005).

The human populations studied are primarily in southern Cameroon. The investigators will continue to focus on several populations of southern Cameroon to gather further information on risk factors for the acquisition of foamy retroviruses following contact with NHPs.

These populations live close to, or in, dense rainforest areas. They are particularly at risk, due to the high biodiversity of NHPs in these regions. The greatest risk comes from relatively frequent contact with NHPs when hunting, which is for both consumption and sale of bushmeat.

OBJECTIVES The project presented herein consists of four phases. These phases can be carried out simultaneously.

Principal objective (phases 1 and 2) The purpose of this work is to carry out a serological and molecular survey to assess the prevalence of foamy virus infection in people at risk of contact with monkeys and to characterize risk factors for interspecies transmission.

This project corresponds to microbiological monitoring and, in particular, the study of the first stages of viral emergence.

Secondary objectives (phases 3 and 4)

1. Investigate possible intrafamilial transmission of foamy viruses from index cases, who all acquired the virus by being bitten by a great ape.
2. Investigate possible biological (especially immuno-virological) and clinical abnormalities in infected individuals through a case-control study. This will require a minimum of 30 index cases and 30 to 60 controls, if possible.

ORGANISATION OF THE STUDY The value and importance of this work on viral emergence will be presented to both administrative and traditional (village chief) local authorities. The investigators will work in three regions of southern Cameroon: the coastal region (Bipindi/Lolodorf/Campo), a more central region (Djoum/Oveng/Mintom/Akonolinga/Somolamo), and in the East in the region of Abong-Mang, Lomié, and Messok.

In these forested areas, the investigators work in Bantu villages (Ngoumba, Fang, Mvae, Zimé, etc.) and with the two different populations of Pygmies, the Bakolas in the West and the Bakas in the East.

Information is provided to each individual and the written consent of all participants collected by physicians.

In Phase 1 of the project, the study is proposed to all adults. There is no selection. A physical examination and blood draw into a 5/10 ml EDTA tube are performed.

In Phase 2, the investigators will specifically search for adults who have been in contact with a NHP during their lifetime. These contacts may include bites, scratches, or other injuries during hunting, or casual encounters with NHPs. An examination and blood draw in a 5/10 ml EDTA tube are performed. The epidemiological data on risk factors are collected through a short questionnaire.

In Phase 3, the investigators will perform a second visit to extend the survey to the nuclear family of infected individuals (spouse and children). An examination and blood draw into a 5/10 ml EDTA tube are performed (Table 1).

During Phase 4, additional clinical and biological examinations will be carried out on infected individuals at the Pasteur Center of Cameroon in Yaoundé (Phase 4). During this visit, saliva is collected. Oral specimens will be collected by rubbing the inside of the cheek with a swab and then rinsing the mouth and collecting the rinse liquid in a sterile bottle. Blood will be collected for further studies. Accommodation in Yaoundé, transportation, and meals of the subjects will be covered by EPVO.

The family study to detect the possible transmission of the virus, and the clinical and biological case-control study, will be carried out during the second phase, if sufficient infected people are detected during the first sero-epidemiological and virological survey.

The EPVO unit at Institut Pasteur is fully responsible for the organization and execution of the field work with logistical support from the IRD (renting a vehicle with driver) and the CPC (reception at the virology laboratory). Prof Antoine Gessain coordinates the project in Paris and Cameroon, and Dr. Edouard Betsem organizes the work in Cameroon.

The samples are aliquoted. Two aliquots of plasma and a peripheral blood buffy coat preparation are frozen at the Pasteur Center in Cameroon. In some cases, peripheral blood mononuclear cells will be obtained on Ficoll and then cultured.

These samples are then sent to the Institut Pasteur in Paris by air, according to current transport standards.

Back in Paris, biological tests and statistical analysis are performed by members of the EPVO unit.

ELIGIBILITY:
Inclusion Criteria:

* Living in a rural zone of Cameroon
* Being > 5 yrs old
* Having received study information and having provided written consent for self and children, if applicable (for all phases)

Exclusion Criteria:

* Having refused to provide consent
* Being less than 5 years old

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The survey has been and will be carried out in villages in southern Cameroon and the target population will change during the four phases of the study as follows:
  1. Initially, all adults encountered (Phase 1).
  2. In the second phase, people who have been in physical contact with monkeys (bites, scratches, wounds, etc.) mainly during hunting and the cleaning of bushmeat
  3. Finally, after screening: focus on infected individuals and inclusion of their immediate family (mainly spouses and children) to study potential intrafamilial transmission (Phase 3).
  4. For infected individuals, an annual clinical, biological and immunological examination, for 3 years (Phase 4). An uninfected person matched for age, sex, ethnic group, and locality will be recruited as a control for each case.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2010-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection with simian foamy virus by determination of the presence of specific antibodies in plasma | 3 years
  Determination of the presence of specific antibodies in plasma through a positive western blot for foamy virus
Infection with simian foamy virus by determination of the presence viral DNA in blood cells | 3 years
  Determination of the presence viral DNA in blood cells through a positive PCR assay using generic amplimers, giving rise to fragments of the integrase gene (425 bp) and LTR (109 bp).

CONTACTS AND LOCATIONS:
Overall Officials: Antoine GESSAIN, MD, Principal Investigator — Institut Pasteur
Locations (1):
- Centre Pasteur du CAmeroun, Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calattini S, Betsem E, Bassot S, Chevalier SA, Mahieux R, Froment A, Gessain A. New strain of human T lymphotropic virus (HTLV) type 3 in a Pygmy from Cameroon with peculiar HTLV serologic results. J Infect Dis. 2009 Feb 15;199(4):561-4. doi: 10.1086/596206. PMID 19099485
- [Background] Calattini S, Betsem EB, Froment A, Mauclere P, Tortevoye P, Schmitt C, Njouom R, Saib A, Gessain A. Simian foamy virus transmission from apes to humans, rural Cameroon. Emerg Infect Dis. 2007 Sep;13(9):1314-20. doi: 10.3201/eid1309.061162. PMID 18252101
- [Background] Calattini S, Chevalier SA, Duprez R, Afonso P, Froment A, Gessain A, Mahieux R. Human T-cell lymphotropic virus type 3: complete nucleotide sequence and characterization of the human tax3 protein. J Virol. 2006 Oct;80(19):9876-88. doi: 10.1128/JVI.00799-06. PMID 16973592
- [Background] Calattini S, Chevalier SA, Duprez R, Bassot S, Froment A, Mahieux R, Gessain A. Discovery of a new human T-cell lymphotropic virus (HTLV-3) in Central Africa. Retrovirology. 2005 May 9;2:30. doi: 10.1186/1742-4690-2-30. PMID 15882466
- [Background] Calattini S, Nerrienet E, Mauclere P, Georges-Courbot MC, Saib A, Gessain A. Natural simian foamy virus infection in wild-caught gorillas, mandrills and drills from Cameroon and Gabon. J Gen Virol. 2004 Nov;85(Pt 11):3313-3317. doi: 10.1099/vir.0.80241-0. PMID 15483245
- [Background] Calattini S, Wanert F, Thierry B, Schmitt C, Bassot S, Saib A, Herrenschmidt N, Gessain A. Modes of transmission and genetic diversity of foamy viruses in a Macaca tonkeana colony. Retrovirology. 2006 Apr 11;3:23. doi: 10.1186/1742-4690-3-23. PMID 16608518
- [Background] Engel G, Hungerford LL, Jones-Engel L, Travis D, Eberle R, Fuentes A, Grant R, Kyes R, Schillaci M. Risk assessment: A model for predicting cross-species transmission of simian foamy virus from macaques (M. fascicularis) to humans at a monkey temple in Bali, Indonesia. Am J Primatol. 2006 Sep;68(9):934-48. doi: 10.1002/ajp.20299. PMID 16900504
- [Background] Gessain A, Mauclere P, Froment A, Biglione M, Le Hesran JY, Tekaia F, Millan J, de The G. Isolation and molecular characterization of a human T-cell lymphotropic virus type II (HTLV-II), subtype B, from a healthy Pygmy living in a remote area of Cameroon: an ancient origin for HTLV-II in Africa. Proc Natl Acad Sci U S A. 1995 Apr 25;92(9):4041-5. doi: 10.1073/pnas.92.9.4041. PMID 7732027
- [Background] Mahieux R, Chappey C, Meertens L, Mauclere P, Lewis J, Gessain A. Molecular characterization and phylogenetic analyses of a new simian T cell lymphotropic virus type 1 in a wild-caught african baboon (Papio anubis) with an indeterminate STLV type 2-like serology. AIDS Res Hum Retroviruses. 2000 Dec 10;16(18):2043-8. doi: 10.1089/088922200750054774. PMID 11153087
- [Background] Mahieux R, Horal P, Mauclere P, Mercereau-Puijalon O, Guillotte M, Meertens L, Murphy E, Gessain A. Human T-cell lymphotropic virus type 1 gag indeterminate western blot patterns in Central Africa: relationship to Plasmodium falciparum infection. J Clin Microbiol. 2000 Nov;38(11):4049-57. doi: 10.1128/JCM.38.11.4049-4057.2000. PMID 11060067
- [Background] Mauclere P, Le Hesran JY, Mahieux R, Salla R, Mfoupouendoun J, Abada ET, Millan J, de The G, Gessain A. Demographic, ethnic, and geographic differences between human T cell lymphotropic virus (HTLV) type I-seropositive carriers and persons with HTLV-I Gag-indeterminate Western blots in Central Africa. J Infect Dis. 1997 Aug;176(2):505-9. doi: 10.1086/514071. PMID 9237719
- [Background] Mauclere P, Mahieux R, Garcia-Calleja JM, Salla R, Tekaia F, Millan J, De The G, Gessain A. A new HTLV type II subtype A isolate in an HIV type 1-infected prostitute from Cameroon, Central Africa. AIDS Res Hum Retroviruses. 1995 Aug;11(8):989-93. doi: 10.1089/aid.1995.11.989. PMID 7492447
- [Background] Meertens L, Mahieux R, Mauclere P, Lewis J, Gessain A. Complete sequence of a novel highly divergent simian T-cell lymphotropic virus from wild-caught red-capped mangabeys (Cercocebus torquatus) from Cameroon: a new primate T-lymphotropic virus type 3 subtype. J Virol. 2002 Jan;76(1):259-68. doi: 10.1128/jvi.76.1.259-268.2002. PMID 11739691
- [Background] Meertens L, Rigoulet J, Mauclere P, Van Beveren M, Chen GM, Diop O, Dubreuil G, Georges-Goubot MC, Berthier JL, Lewis J, Gessain A. Molecular and phylogenetic analyses of 16 novel simian T cell leukemia virus type 1 from Africa: close relationship of STLV-1 from Allenopithecus nigroviridis to HTLV-1 subtype B strains. Virology. 2001 Sep 1;287(2):275-85. doi: 10.1006/viro.2001.1018. PMID 11531406
- [Background] Meertens L, Shanmugam V, Gessain A, Beer BE, Tooze Z, Heneine W, Switzer WM. A novel, divergent simian T-cell lymphotropic virus type 3 in a wild-caught red-capped mangabey (Cercocebus torquatus torquatus) from Nigeria. J Gen Virol. 2003 Oct;84(Pt 10):2723-2727. doi: 10.1099/vir.0.19253-0. PMID 13679606
- [Background] Nerrienet E, Meertens L, Kfutwah A, Foupouapouognigni Y, Ayouba A, Gessain A. Simian T cell leukaemia virus type I subtype B in a wild-caught gorilla (Gorilla gorilla gorilla) and chimpanzee (Pan troglodytes vellerosus) from Cameroon. J Gen Virol. 2004 Jan;85(Pt 1):25-29. doi: 10.1099/vir.0.19314-0. PMID 14718616
- [Background] Nerrienet E, Meertens L, Kfutwah A, Foupouapouognigni Y, Gessain A. Molecular epidemiology of simian T-lymphotropic virus (STLV) in wild-caught monkeys and apes from Cameroon: a new STLV-1, related to human T-lymphotropic virus subtype F, in a Cercocebus agilis. J Gen Virol. 2001 Dec;82(Pt 12):2973-2977. doi: 10.1099/0022-1317-82-12-2973. PMID 11714973
- [Background] Switzer WM, Salemi M, Shanmugam V, Gao F, Cong ME, Kuiken C, Bhullar V, Beer BE, Vallet D, Gautier-Hion A, Tooze Z, Villinger F, Holmes EC, Heneine W. Ancient co-speciation of simian foamy viruses and primates. Nature. 2005 Mar 17;434(7031):376-80. doi: 10.1038/nature03341. PMID 15772660
- [Background] Wolfe ND, Switzer WM, Carr JK, Bhullar VB, Shanmugam V, Tamoufe U, Prosser AT, Torimiro JN, Wright A, Mpoudi-Ngole E, McCutchan FE, Birx DL, Folks TM, Burke DS, Heneine W. Naturally acquired simian retrovirus infections in central African hunters. Lancet. 2004 Mar 20;363(9413):932-7. doi: 10.1016/S0140-6736(04)15787-5. PMID 15043960
- [Derived] Dynesen LT, Fernandez I, Coquin Y, Delaplace M, Montange T, Njouom R, Bilounga-Ndongo C, Rey FA, Gessain A, Backovic M, Buseyne F. Neutralization of zoonotic retroviruses by human antibodies: Genotype-specific epitopes within the receptor-binding domain from simian foamy virus. PLoS Pathog. 2023 Apr 24;19(4):e1011339. doi: 10.1371/journal.ppat.1011339. eCollection 2023 Apr. PMID 37093892
- [Derived] Couteaudier M, Montange T, Njouom R, Bilounga-Ndongo C, Gessain A, Buseyne F. Plasma antibodies from humans infected with zoonotic simian foamy virus do not inhibit cell-to-cell transmission of the virus despite binding to the surface of infected cells. PLoS Pathog. 2022 May 23;18(5):e1010470. doi: 10.1371/journal.ppat.1010470. eCollection 2022 May. PMID 35605011
- [Derived] Buseyne F, Betsem E, Montange T, Njouom R, Bilounga Ndongo C, Hermine O, Gessain A. Clinical Signs and Blood Test Results Among Humans Infected With Zoonotic Simian Foamy Virus: A Case-Control Study. J Infect Dis. 2018 Jun 5;218(1):144-151. doi: 10.1093/infdis/jiy181. PMID 29608711